CLINICAL TRIAL: NCT01814202
Title: A Double-blind, Randomized, Placebo-controlled Clinical Trial (Pilot Phase) to Evaluate the Efficacy of a Medical Nutrition Product, PTM202, in Children With Acute Diarrhea
Brief Title: Study With Medical Nutrition Product PTM202 in Pediatric Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PanTheryx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTM.2012.002; PR-13002 (Other: icddr,b)
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Acute Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTM202 (Experimental): PTM202 is a medical nutrition product
  Interventions: Other: PTM202
- Placebo (Placebo Comparator): The placebo is a placebo for PTM202, a food product that can not be distinguished from PTM202 by appearance, taste or odor
  Interventions: Other: Placebo

INTERVENTIONS:
Other: PTM202
  Arms: PTM202
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a medical nutrition product, PTM202, along with standard of care, enhances recovery and reduces diarrhea morbidity in young children

ELIGIBILITY:
Inclusion Criteria:

* males or females between 6 months and 5 years of age
* acute diarrhea (<48 hours) without interfering co-morbidities
* guardian willing to have child admitted to hospital as an inpatient for 96 hours and to return to the clinic with the child on Day 7 for a final evaluation
* Guardian is willing and able to report to the Investigator information on stool frequency, stool consistency and food and water intakes during the follow up phase.
* Written informed consent must be obtained prior to admission to this study.
* The subject has a physical examination that reveals no clinically significant abnormalities other than those expected for subjects with acute infectious diarrhea.

Exclusion Criteria:

* Suspected or confirmed cholera
* Suspected dysentery
* Symptom duration >48 hours at screening
* Vomiting severity that is like to make administration and retention of test article impossible
* Severe malnutrition (defined as weight for height of less than -3 SD below median, per WHO Standards (6).
* Child already receiving antibiotics or anti-motility drugs for this diarrhea episode prior to screening.
* History of hypersensitivity or allergy to milk or egg

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
diarrhea duration | 7 days

SECONDARY OUTCOMES:
food intake | 7 days
stool frequency | 7 days
stool consistency | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Shafiqul A Sarker, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Dhaka Division, Bangladesh